CLINICAL TRIAL: NCT04042584
Title: Pre-hospital Optimization of Triage of Stroke Suspicions: Bringing an Embedded Visio Conference Device
Brief Title: Visio-conference for Pre-hospital Triage of Stroke Suspicions
Acronym: OPTIC-AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/42
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Cerebrovascular Disorders
Keywords: Stroke; Mechanical thrombectomy; Tele-evaluation; Emergency medical service; Pre hospital
MeSH Terms: conditions — Stroke; Ischemic Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visio conference device evaluation (Experimental): Neurological tele-evaluation by a neurologist
  Interventions: Procedure: Visio conference device evaluation (DVCM)

INTERVENTIONS:
Procedure: Visio conference device evaluation (DVCM) — Standard neurological tele-evaluation (limited to 15minutes) remotely carried out by a first neurologist via a tablet (DVCM) and an operator. A second neurologist assist at the assessment without intervention next to the patient. Once the remote assessment is complet, the second neurologist ensure the continuation of standard patient care.

SUMMARY:
Interventionnal Study to investigate the accuracy of our clinical based algorithm performed by using a visioconference device to assess the eligibility of acute recanalisation treatment (intraveinous thrombolysis (IVT) and/or mechanical thrombectomie (TM). Clinical identification of type of treatment is needed is pre-hospital triage of these patients.

DETAILED DESCRIPTION:
The outcome of ischemic stroke (IS) with large artery occlusion (LVO) is related to the volume of infarcted brain witch is related to the delay of arterial recanalisation. IVT is available in multiple stroke units in France but, in case of LVO, the association with TM is needed. The availability of endovascular capable centers is limited to tertiary care hospitals. As a result, pre-hospital identification of these patients is a priority and the optimization of the triage can be done by a clinical algorithm carried out by a neurological tele-evaluation.

OPTIC-AVC is a multi-phase study. This phase is about the evaluation of accuracy of our algorithm performed by a quick and standardized neurological tele-evaluation to predict the eligibility for recanalisation treatment (IVT and/or TM) of patients suspected of acute stroke in the emergency setting. The effective therapeutic decision for each patient, performed by another neurologist, will be blind to the theoretical therapeutic decision resulting from the algorithm.

Theoretical and effective therapeutic decision will be compared a posteriori

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Suspicion of acute symptomatic stroke whose first symptoms are less than 24 hours old
* Free Consent, informed writing signed by the participant or the person of confidence and the investigator (no later than the day of inclusion and before any examination required by research)

Exclusion Criteria:

* Stupor or coma requiring orotracheal intubation
* Rankin pre stroke > 4
* Severe cognitive impairement
* Contraindication to the realiszation of angiographic imaging
* Participation refusal
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Final effective therapeutic decision | Day 0
  Thrombolysis and/or thrombectomy : yes/no

SECONDARY OUTCOMES:
Therapeutic conviction | Day 0
  Theoretical conviction using Likert scales between the neurologist at the patient bedside and the neurologist using the device for tele-evaluation
Remote evaluation failure | Day 0
  Remote evaluation failure rate
Theoretical therapeutic decision | Day 0
  Theoretical therapeutic decision of the algorithm : thrombolysis and/or thrombectomy [yes/no]

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France